CLINICAL TRIAL: NCT02588261
Title: An Open-label, Randomized Phase 3 Efficacy Study of ASP8273 vs Erlotinib or Gefitinib in First-line Treatment of Patients With Stage IIIB/IV Non-small Cell Lung Cancer Tumors With EGFR Activating Mutations
Brief Title: A Study of ASP8273 vs. Erlotinib or Gefitinib in First-line Treatment of Patients With Stage IIIB/IV Non-small Cell Lung Cancer Tumors With EGFR Activating Mutations
Acronym: SOLAR
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Following recommendation by SOLAR Study IDMC, Astellas closed enrollment in ASP8273 studies
Sponsor: Astellas Pharma Global Development, Inc. (Industry)
Responsible Party: Sponsor
Organization: Astellas Pharma Inc (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 8273-CL-0302; 2015-002894-39 (EudraCT Number)
Record Dates: First submitted 2015-10-26; First posted 2015-10-27 (Estimated); Results first posted 2019-02-12 (Actual); Last update posted 2024-12-10 (Actual); Status verified 2024-11

CONDITIONS: Non-small Cell Lung Cancer (NSCLC)
Keywords: erlotinib; EGFR mutation; naquotinib; Non-small cell lung cancer (NSCLC); ASP8273; gefitinib
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — naquotinib; Erlotinib Hydrochloride; Gefitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- ASP8273 (Experimental): Participants received 300 mg of ASP8273 orally once daily in 28-day cycles until one of the discontinuation criteria was met (developed radiological progressive disease, required to receive local or systemic anti-cancer treatment, developed unacceptable toxicity, participant pregnancy, investigator decision, required to receive significant surgical procedure, participant protocol deviation or noncompliance, participant decline of further treatment and participant lost to follow-up).
  Interventions: Drug: naquotinib mesilate
- erlotinib or gefitinib (Active Comparator): Participants received 150 mg of erlotinib or 250 mg of gefitinib orally once daily in 28-day cycles until one of the discontinuation criteria was met (developed radiological progressive disease, required to receive local or systemic anti-cancer treatment, developed unacceptable toxicity, participant pregnancy, investigator decision, required to receive significant surgical procedure, participant protocol deviation or noncompliance, participant decline of further treatment and participant lost to follow-up).
  Interventions: Drug: Erlotinib; Drug: Gefitinib

INTERVENTIONS:
Drug: naquotinib mesilate — Participants received ASP8273 300 mg orally once daily on an empty stomach (no food for at least 2 hours before and 1 hour after taking drug) at approximately the same time every day.
  Other Names: ASP8273
  Arms: ASP8273
Drug: Erlotinib — Participants received erlotinib 150 mg orally once daily on an empty stomach (no food for at least 2 hours before and 1 hour after taking drug) at approximately the same time every day. At the beginning of the trial, prior to site initiation and shipment of study drug supplies, each investigator selected either erlotinib or gefitinib to be utilized for all participants randomized to the comparator arm at their site.
  Other Names: Tarceva; OSI-774
  Arms: erlotinib or gefitinib
Drug: Gefitinib — Participants received gefitinib 250 mg was taken orally once daily with water, with or without food, at approximately the same time every day. At the beginning of the trial, prior to site initiation and shipment of study drug supplies, each investigator selected either erlotinib or gefitinib to be utilized for all participants randomized to the comparator arm at their site.
  Arms: erlotinib or gefitinib

SUMMARY:
The purpose of the study was to evaluate the progression free survival (PFS), based on independent radiologic review (IRR), of ASP8273 compared to erlotinib or gefitinib in patients with locally advanced, metastatic or unresectable stage IIIB/IV adenocarcinoma non-small cell lung cancer (NSCLC) with epidermal growth factor receptor (EGFR) activating mutations.

This study also assessed Overall survival (OS); Overall response rate (ORR) as assessed by IRR; PFS as assessed by the investigator; Disease control rate (DCR) as assessed by IRR; Duration of Response (DOR) by IRR; Safety of ASP8273; and Quality of Life (QOL) and patient-reported outcome (PRO) parameters.

ELIGIBILITY:
Inclusion Criteria:

* Subject agrees not to participate in another interventional study while on treatment.
* Female subject must either:

  * Be of nonchildbearing potential: postmenopausal (defined as at least 1 year without any menses) prior to Screening, or documented surgically sterile
  * Or, if of childbearing potential: Agree not to try to become pregnant during the study and for 28 days after the final study drug administration; And have a negative serum pregnancy test at Screening; And, if heterosexually active, agree to consistently use 2 forms of highly effective birth control (at least 1 of which must be a highly effective method and one must be a barrier method) starting at Screening and throughout the study period and for 28 days after the final study drug administration.
* Female subject must not be breastfeeding at Screening or during the study period, and for 28 days after the final study drug administration.
* Female subject must not donate ova starting at Screening and throughout the study period, and for 28 days after the final study drug administration.
* Male subject and their female spouse/partners who are of childbearing potential must be using highly effective contraception consisting of 2 forms of birth control (1 of which must be a barrier method) starting at Screening and continue throughout the study period and for 90 days after the final study drug administration.
* Male subject must not donate sperm starting at Screening and throughout the study period and for 90 days after the final study drug administration.
* Subject has Eastern Cooperative Oncology Group (ECOG) performance status ≤ 2.
* Subject has histologically confirmed locally advanced, metastatic or unresectable Stage IIIB/IV adenocarcinoma NSCLC (newly diagnosed or recurrent). Subjects with mixed histology are eligible if adenocarcinoma is the predominant histology.
* Subject has predicted life expectancy ≥ 12 weeks in the opinion of the investigator.
* Subject must meet all of the following criteria on the laboratory tests that will be analyzed centrally within 7 days prior to the first dose of study drug. In case of multiple laboratory data within this period, the most recent data should be used.

  * Neutrophil count > 1,000/mm3
  * Platelet count ≥ 7.5 x 104 /mm3
  * Hemoglobin > 8.0 g/dL
  * Serum creatinine ˂ 2.0 x upper limit of normal (ULN) or an estimated glomerular filtration rate (eGFR) of > 50 mL/min as calculated by the Cockcroft Gault Method
  * Total bilirubin ˂1.5 x ULN (except for subjects with documented Gilbert's syndrome)
  * AST and ALT ˂ 3.0 x ULN or ≤ 5 x ULN if subject has documented liver metastases
  * Serum sodium level is ≥ 130 mmol/L
* Subject has an EGFR activating mutation (exon 19 deletion or exon 21 L858R), with or without T790M mutation, by local or central testing on examination of a NSCLC FFPE specimen (archival or fresh biopsy). Subjects harboring both exon 19 deletion and exon 21 L858R mutations are not eligible. A tissue sample from the same block used to determine eligibility by local testing should be available to send to the central lab for confirmatory testing. Subjects randomized based on local results indicating presence of EGFR mutation may remain on study if central results are discordant.
* Subject must have at least 1 measureable lesion based on RECIST V1.1. Previously irradiated lesions will not be considered as measurable lesions.

Exclusion Criteria:

* Subject has received intervening anticancer treatment or previous treatment with chemotherapy for metastatic disease other than palliative local radiation to painful bone metastases completed at least 1 week prior to the first dose of study drug. The administration of neoadjuvant or adjuvant chemotherapy is allowed as long as it has finalized ≥ 6 months before the first dose of study drug.
* Subject has received a prior treatment with a therapeutic agent targeting EGFR (e.g., afatinib, dacomitinib, ASP8273, etc).
* Subject has received investigational therapy within 28 days or 5 half-lives prior to the first dose of study drug.
* Subject has received radiotherapy within 1 week prior to the first dose of study drug. If the subject received radiotherapy > 1 week prior to study treatment, the irradiated lesion cannot be the only lesion used for evaluating response.
* Subject has symptomatic central nervous system (CNS) metastasis. Subject with previously treated brain or CNS metastases are eligible provided that the subject has recovered from any acute effects of radiotherapy, does not have brain metastasis related symptoms, is not requiring systemic steroids for at least 2 weeks prior to study drug administration, and any whole brain radiation therapy was completed at least 4 weeks prior to study drug administration, or any stereotactic radiosurgery (SRS) was completed at least 2 weeks prior to study drug administration. Steroid inhaler use or ointment treatment for other concomitant medical disease is permitted.
* Subject has received blood transfusions or hematopoietic factor therapy within 14 days prior to the first dose of study drug.
* Subject has had a major surgical procedure (other than a biopsy) within 14 days prior to the first dose of study drug, or one is planned during the course of the study.
* Subject has a known history of a positive test for human immunodeficiency virus (HIV) infection.
* Subject has known history of serious hypersensitivity reaction to a known ingredient of ASP8273, erlotinib or gefitinib.
* Subject has evidence of an active infection requiring systemic therapy within 14 days prior to the planned first dose of study drug.
* Subject has severe or uncontrolled systemic diseases including uncontrolled hypertension (blood pressure > 150/100 mmHg) or active bleeding diatheses.
* Subject has history of drug-induced interstitial lung disease (ILD) or any evidence of active ILD.
* Subject has ongoing cardiac arrhythmia that is Grade ≥ 2 or uncontrolled atrial fibrillation of any grade.
* Subject currently has Class 3 or 4 New York Heart Association congestive heart failure.
* Subject has history of severe/unstable angina, myocardial infarction or cerebrovascular accident within 6 months prior to the planned first dose of study drug.
* Subject has history of gastrointestinal ulcer or gastrointestinal bleeding within 3 months prior to the planned first dose of study drug.
* Subject has concurrent corneal disorder or any ophthalmologic condition which, in the investigator's opinion, makes the subject unsuitable for study participation (i.e., advanced cataracts, glaucoma).
* Subject has difficulty taking oral medication or any digestive tract dysfunction or inflammatory bowel disease that would interfere with the intestinal absorption of drug.
* Subject has another past or active malignancy which requires treatment. Prior carcinoma in situ or non-melanoma skin cancer after curative resection are permitted.
* Subject has any condition which, in the investigator's opinion, makes the subject unsuitable for study participation.
* Subject has received potent CYP 3A4 inhibitors within 7 days prior to first dose of study drug or proton pump inhibitors such as omeprazole within 14 days prior to first dose of study drug.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 530 (Actual)
Dates: Start 2016-02-11 (Actual); Primary Completion 2017-12-21 (Actual); Study Completion 2017-12-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Astellas Pharma Global Development, Inc.
Locations (167):
- United States (25):
  - Site US10029, Beverly Hills, California
  - Site US10025, Fountain Valley, California
  - Site US10036, La Jolla, California
  - Site US10051, Loma Linda, California
  - Site US10033, Los Angeles, California
  - Site US10031, Oxnard, California
  - Site US10052, Redondo Beach, California
  - Site US10003, Santa Monica, California
  - Site US10018, Whittier, California
  - Site US10047, Glenwood Springs, Colorado
  - Site US10013, Aventura, Florida
  - Site US10048, St. Petersburg, Florida
  - Site US10050, Atlanta, Georgia
  - Site US10042, Baton Rouge, Louisiana
  - Site US10037, Scarborough, Maine
  - Site US10034, Boston, Massachusetts
  - Site US10030, Minneapolis, Minnesota
  - Site US10027, Rochester, Minnesota
  - Site US10045, Albuquerque, New Mexico
  - Site US10012, Mount Kisco, New York
  - Site US10021, Bethlehem, Pennsylvania
  - Site US10009, Nashville, Tennessee
  - Site US10023, Nashville, Tennessee
  - Site US10011, Lacey, Washington
  - Site US10046, Milwaukee, Wisconsin
- Australia (6):
  - Site AU61003, Randwick, New South Wales
  - Site AU61007, Woolloongabba, Queensland
  - Site AU61005, Adelaide, South Australia
  - Site AU61008, East Melbourne, Victoria
  - Site AU61002, Fitzroy, Victoria
  - Site AU61004, Footscray, Victoria
- Site BE32002, Ghent, West-Vlaanderen, Belgium
- Canada (2):
  - Site CA15006, Toronto, Ontario
  - Site CA15002, Montreal, Quebec
- Chile (3):
  - Site CL56002, Viña del Mar, Región de Valparaíso
  - Site CL56007, Viña del Mar, Región de Valparaíso
  - Site CL56001, Santiago, Región Metropolitana de Santia
- France (8):
  - Site FR33010, Pessac, Gironde
  - Site FR33011, Suresnes, Hauts-de-Seine
  - Site FR33003, Créteil, Ilej-de-France
  - Site FR33004, Tours, Indre-et-Loire
  - Site FR33006, Grenoble, Isère
  - Site FR33009, Saint Priest En Jarez, Pays de la Loire Region
  - Site FR33012, Bayonne, Pyrénées-Atlantiques
  - Site FR33007, Pierre-Bénite, Rhône
- Germany (6):
  - Site DE49008, Freiburg im Breisgau, Baden-Wurttemberg
  - Site DE49005, Karlsruhe, Baden-Wurttemberg
  - Site DE49003, Gauting, Bavaria
  - Site DE49006, Würzburg, Bavaria
  - Site DE49007, Kassel, Hesse
  - Site DE49004, Cologne, North Rhine-Westphalia
- Hungary (6):
  - Site HU36002, Székesfehérvár, Fejér
  - Site HU36003, Tatabánya, Tatabánya
  - Site HU36006, Szombathely, Vas County
  - Site HU36004, Farkasgyepű, Veszprém megye
  - Site HU36007, Budapest
  - Site HU36001, Budapest
- Italy (10):
  - Site IT39004, Monza, Lombardy
  - Site IT39009, Rozzano, Lombardy
  - Site IT39011, Aviano, Pordenone
  - Site IT39003, Bergamo
  - Site IT39015, Brescia
  - Site IT39002, Cremona
  - Site IT39013, Lucca
  - Site IT39014, Milan
  - Site IT39012, Piacenza
  - Site IT39008, Roma
- Japan (21):
  - Site JP81018, Matsuyama, Ehime
  - Site JP81013, Hiroshima, Hirosima [Hiroshima]
  - Site JP81014, Sapporo, Hokkaidô
  - Site JP81017, Osakasayama-shi, Hukuoka [Fukuoka]
  - Site JP81008, Kurume, Hukuoka
  - Site JP81024, Kobe, Hyōgo
  - Site JP81015, Kanazawa, Isikawa [Ishikawa]
  - Site JP81010, Yokohama, Kanagawa
  - Site JP81025, Yokohama, Kanagawa
  - Site JP81012, Sendai, Miyagi
  - Site JP81016, Kurashiki, Okayama-ken
  - Site JP81005, Miyakojima-ku, Osaka
  - Site JP81020, Osakasayama-shi, Osaka
  - Site JP81019, Sunto-gun, Shizuoka
  - Site JP81001, Sunto-gun, Sizuoka [Shizuoka]
  - Site JP81004, Tokyo, Tôkyô [Tokyo]
  - Site JP81022, Niigata
  - Site JP81006, Okayama
  - Site JP81023, Wakayama
  - Site JP81021, Hirakata, Ôsaka [Osaka]
  - Site JP81002, Ōsaka-sayama, Ôsaka [Osaka]
- Malaysia (3):
  - Site MY60001, Kuantan Pahang, Pahang
  - Site MY60002, George Town, Pulau Pinang
  - Site MY60004, Kuching, Sarawak
- Netherlands (2):
  - Site NL31001, Arnhem, Gelderland
  - Site NL31006, Alkmaar, North Holland
- Peru (3):
  - Site PE51001, Cercado de Lima, Arequipa
  - Site PE51008, Miraflores, Lima region
  - Site PE51004, San Isidro, Lima region
- Portugal (4):
  - Site PT35101, Amadora, Lisbon District
  - Site PT35104, Lisbon, Lisbon District
  - Site PT35103, Coimbra
  - Site PT35102, Lisbon
- Romania (7):
  - Site RO40004, Floreşti, Cluj
  - Site RO40001, Craiova, Dolj
  - Site RO40010, Craiova, Dolj
  - Site RO40007, Ploieşti, Prahova
  - Site RO40008, Timișoara, Timiș County
  - Site RO40012, Bucharest
  - Site RO40006, Sibiu
- Russia (6):
  - Site RU70012, Arkhangelsk, Arkhangelskaya oblast
  - Site RU70017, Ufa, Bashkortostan Republic
  - Site RU70009, Magnitogorsk, Chelyabinsk Oblast
  - Site RU70016, Nal'chik, Kabardino-Balkarskaya Respublika
  - Site RU70008, Pyatigorsk, Stavropol Kray
  - Site RU70001, Saint Petersburg
- Singapore (2):
  - Site SG65001, Singapore, Central Singapore
  - Site SG65002, Singapore, Central Singapore
- South Korea (16):
  - Site KR82010, Busan Gwang'yeogsi, Busan Gwang'yeogsi
  - Site KR82004, Suwon, Gyeonggi-do
  - Site KR82016, Suwon, Gyeonggido [Kyonggi-do]
  - Site KR82017, Bundang, Gyeonggido
  - Site KR82009, Jinju, Gyeongsangnam-do
  - Site KR82003, Jeonju, Jeonrabugdo[Chollabuk-do]
  - Site KR82005, Cheongiu, North Chungcheong
  - Site KR82002, Seoul, Seoul Teugbyeolsi [Seoul-T'ukp]
  - Site KR82001, Seoul, Seoul Teugbyeolsi [Seoul-T'ukp]
  - Site KR82013, Seoul, Seoul Teugbyeolsi [Seoul-T'ukp]
  - Site KR82007, Seoul, Seoul Teugbyeolsi [Seoul-T'ukp]
  - Site KR82008, Seoul, Seoul Teugbyeolsi [Seoul-T'ukp]
  - Site KR82006, Seoul, Seoul Teugbyeolsi [Seoul-T'ukp]
  - Site KR82015, Seoul, Seoul Teugbyeolsi [Seoul-T'ukp]
  - Site KR82014, Seoul, Seoul Teugbyeolsi
  - Site KR82011, Ulsan, Ulsan Gwang'yeogsi
- Spain (10):
  - Site ES34003, Barcelona, Catalonia
  - Site ES34008, San Sebastian, Guipuzcoa, Guipúzcoa
  - Site ES34010, Málaga, Málaga
  - Site ES34006, Madrid
  - Site ES34016, Madrid
  - Site ES34004, Ourense
  - Site ES34005, Seville
  - Site ES34015, Valencia
  - Site ES34017, Valencia
  - Site ES34002, Valencia
- Taiwan (9):
  - Site TW88605, Taichung, Taichung
  - Site TW88607, Taoyuan Hsien, Taoyuan
  - Site TW88606, Kaohsiung City
  - Site TW88603, Taichung
  - Site TW88601, Tainan
  - Site TW88604, Tainan
  - Site TW88608, Taipei
  - Site TW88609, Taipei
  - Site TW88611, Taipei
- Thailand (6):
  - Site TH66011, Chom Thong, Chiang Mai
  - Site TH66001, Bangkok, Krung Thep Maha Nakhon [Bangkok]
  - Site TH66012, Bangkok, Krung Thep Maha Nakhon [Bangkok]
  - Site TH66002, Chiang Rai
  - Site TH66004, Khon Kaen
  - Site TH66006, Songkhla
- Ukraine (8):
  - Site UA38006, Chernivtsi, Chernivtsi Oblast
  - Site UA38001, Dnipropetrovsk, Dnipropetrovsk Oblast
  - Site UA38005, Kryvyi Rih, Dnipropetrovsk Oblast
  - Site UA38008, Ivano-Frankivsk, Ivano-Frankivsk Oblast
  - Site UA38004, Lviv, Lviv Oblast
  - Site UA38007, Lutsk, Volyn Oblast
  - Site UA38009, Uzhhorod, Zakarpattia Oblast
  - Site UA38003, Uzhhorod, Zakarpattia Oblast
- United Kingdom (3):
  - Site GB44002, Middlesex, Hertfordshire
  - Site GB44001, Liverpool, Wirral
  - Site GB44003, Sheffield

IPD SHARING:
Plan to Share IPD: Yes
Access to anonymized individual participant level data collected during the study, in addition to study-related supporting documentation, is planned for studies conducted with approved product indications and formulations, as well as products terminated during development. Studies conducted with product indications or formulations that remain active in development are assessed after study completion to determine if Individual Participant Data can be shared. Further details on Astellas' data sharing policy can be found at https://www.clinicaltrials.astellas.com/transparency/.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Access to participant level data is offered to researchers after publication of the primary manuscript (if applicable) and is available as long as Astellas has legal authority to provide the data..
Access Criteria: Researchers must submit a proposal to conduct a scientifically relevant analysis of the study data. The research proposal is reviewed by an Independent Research Panel. If the proposal is approved, access to the study data is provided in a secure data sharing environment after receipt of a signed Data Sharing Agreement.
URL: https://www.clinicaltrials.astellas.com/transparency/

REFERENCES:
- [Derived] Kelly RJ, Shepherd FA, Krivoshik A, Jie F, Horn L. A phase III, randomized, open-label study of ASP8273 versus erlotinib or gefitinib in patients with advanced stage IIIB/IV non-small-cell lung cancer. Ann Oncol. 2019 Jul 1;30(7):1127-1133. doi: 10.1093/annonc/mdz128. PMID 31070709
- See also: Link to results on the Astellas Clinical Study Results website — https://astellasclinicalstudyresults.com/hcp/study.aspx?ID=293

RESULTS

PARTICIPANT FLOW:
Recruitment Details: First-line participants with locally advanced, metastatic or unresectable stage IIIB/IV adenocarcinoma NSCLC with EGFR activating mutation (exon 19 deletion or exon 21 L858R) with or without a T790M mutation who had not previously been treated with an EGFR inhibitors were enrolled in 201 sites in 23 countries.
Pre-assignment Details: Eligible participants were stratified according to the following: Eastern Cooperative Oncology Group (ECOG) performance status (0, 1 or 2), Epidermal growth factor receptor (EGFR) mutation status (exon 19 deletion or mutations in exon 21 [L858R]), Tyrosine kinase inhibitor (TKI) chosen (erlotinib or gefitinib) and race (Asian versus non-Asian).
Period: Overall Study
Arm/Group | ASP8273 | Erlotinib or Gefitinib
Started | 267 | 263
Treated | 265 | 262
Completed | 0 | 0
Not Completed | 267 | 263
Not completed — Study Terminated by Sponsor | 157 | 142
Not completed — Protocol Deviation | 1 | 0
Not completed — Death | 1 | 2
Not completed — Withdrawal by Subject | 12 | 8
Not completed — Noncompliance with Study Drug | 0 | 1
Not completed — Miscellaneous | 5 | 4
Not completed — Progressive Disease | 61 | 82
Not completed — Adverse Event | 29 | 24
Not completed — Lost to Follow-up | 1 | 0

BASELINE CHARACTERISTICS:
Population: The analysis population for all baseline measures consisted of all participants who were randomized in the study.
Groups:
- Total: Total of all reporting groups
Arm/Group | ASP8273 | Erlotinib or Gefitinib | Total
Number analyzed (Participants) | 267 | 263 | 530
Age, Continuous [Mean (Standard Deviation); unit: Years] | 66.6 (10.6) | 65.0 (11.5) | 65.8 (11.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 171 | 153 | 324
  Male | 96 | 110 | 206
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 12 | 11 | 23
  Not Hispanic or Latino | 244 | 245 | 489
  Unknown or Not Reported | 11 | 7 | 18
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 89 | 88 | 177
  Black or African American | 3 | 0 | 3
  Asian | 162 | 163 | 325
  American Indian or Alaska Native | 3 | 1 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Other | 1 | 3 | 4
  Missing | 9 | 8 | 17
Investigator Prerandomization Selected TKI at Randomization [Count of Participants; unit: Participants]
  Erlotinib | 153 | 151 | 304
  Gefitinib | 114 | 112 | 226
ECOG Performance Status at Randomization [Count of Participants; unit: Participants] — ECOG Performance Status is composed of 6 grades: 0 - Fully active, able to carry on all predisease performance without restriction; 1 - Restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature; 2 - Ambulatory and capable of all self-care but unable to carry out any work activities, Up and about more than 50% of waking hours; 3 - Capable of only limited self-care, confined to bed or chair more than 50% of waking hours; 4 - Completely disabled, Cannot carry on any self-care, Totally confined to bed or chair; 5 - Dead.
  Participants
    Grade 0 | 103 | 103 | 206
    Grade 1 | 155 | 152 | 307
    Grade 2 | 9 | 8 | 17
EGFR Mutation Status at Randomization [Count of Participants; unit: Participants]
  Exon 19 Deletion | 149 | 147 | 296
  Exon 21 L858R | 118 | 116 | 234
Race (Asian vs Non-Asian) at Randomization [Count of Participants; unit: Participants]
  Asian | 163 | 162 | 325
  Non-Asian | 104 | 101 | 205

OUTCOME MEASURES:

1. Primary Outcome: Progression Free Survival (PFS) as Assessed by Independent Radiologic Review (IRR)
Description: PFS was defined as the time from the date of randomization until the date of radiological disease progression or until death due to any cause, based on the Response Evaluation Criteria in Solid Tumors (RECIST) v1.1, as assessed by IRR. Results are based Kaplan-Meier estimate. If a participant had neither progressed nor died, who received any further anticancer therapy for the disease before radiological progression, the participant was censored at the date of last radiological assessment. If progression or death occurred after missing 2 scheduled radiological assessments, the participant was censored at the date of last radiological assessment or at the date of randomization if no post-baseline radiological assessment was available.
Time Frame: From date of randomization up to data cut-off date 09 May 2017 (approximately 15 months)
Population: The analysis population was the full analysis set (FAS), which consisted of all participants who were randomized.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | ASP8273 | Erlotinib or Gefitinib
Number analyzed (Participants) | 267 | 263
months | 9.26 [5.62 to 11.07] | 9.59 [8.77 to NA] — Data could not be calculated due to low number of events.
Statistical Analysis 1: Comparison: ASP8273 vs Erlotinib or Gefitinib; Comparison between ASP8273 and Erlotinib or Gefitinib treatment groups was performed using log-rank test stratified by ECOG (0 and 1 vs 2), EGFR mutation type (exon 19 deletion or exon 21 L858R) and TKI chosen by the site (erlotinib or gefitinib) before randomization. Comparison was tested at 1-sided significance level of 0.025. Hazard ratio based on Cox proportional hazards model. Assuming proportional hazards, HR < 1 indicated a reduction in hazard rate in favor of ASP8273 treatment group; Test type: Superiority; p = 0.992, Log Rank; Hazard Ratio (HR) = 1.611, 95% CI 2-sided [1.086 to 2.391]

2. Secondary Outcome: Percentage of Deaths
Description: All events of death after the first study drug administration were included.
Time Frame: From date of randomization up to data cut-off date 21 Dec 2017 (approximately 22 months)
Population: The analysis population was the safety analysis set (SAF), which consisted of all participants who took at least one dose of study drug.
Measure: Number; unit: percentage of participants
Arm/Group | ASP8273 | Erlotinib or Gefitinib
Number analyzed (Participants) | 265 | 262
percentage of participants | 14.7 | 13.4

3. Secondary Outcome: Percentage of Participants With Objective Response (OR)
Description: Percentage of participants with OR was defined as the proportion of participants with best overall response as complete response (CR) or partial response (PR) without confirmation based on the RECIST v1.1 as assessed by the blinded IRR. CR was defined as disappearance of all target and nontarget lesions. Any pathological lymph nodes (whether target or nontarget) must have reduction in short axis to < 10 mm from baseline measurement. PR was defined as at least a 30% decrease in the sum of diameters (longest for nonnodal lesions, short axis for nodal lesions) of target lesions taking as reference to the baseline sum of diameters.
Time Frame: From date of first dose of study drug up to data cut-off date 09 May 2017 (approximately 15 months)
Population: The analysis population was the FAS.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | ASP8273 | Erlotinib or Gefitinib
Number analyzed (Participants) | 267 | 263
percentage of participants | 33.0 [27.4 to 39.0] | 47.9 [41.7 to 54.1]
Statistical Analysis 1: Comparison: ASP8273 vs Erlotinib or Gefitinib; Comparison between ASP8273 and Erlotinib or Gefitinib treatment groups was performed using stratified Cochran-Mantel-Haenszel (CMH) test, stratified by ECOG (0 and 1 vs 2), EGFR mutation type (exon 19 deletion or exon 21 L858R) and TKI chosen by the site (erlotinib or gefitinib) before randomization. Comparison was tested at 1-sided significance level of 0.025; Test type: Superiority; p = 1.000, Cochran-Mantel-Haenszel

4. Secondary Outcome: PFS as Assessed by the Investigator
Description: PFS was defined as the time from the date of randomization until the date of radiological disease progression or until death due to any cause, based on RECIST V1.1, as assessed by local investigator. Results are based Kaplan-Meier estimate. If a participant had neither progressed nor died, who received any further anticancer therapy for the disease before radiological progression, the participant was censored at the date of last radiological assessment. If progression or death occurred after missing 2 scheduled radiological assessments, the participant was censored at the date of last radiological assessment or at the date of randomization if no post-baseline radiological assessment was available.
Time Frame: From date of randomization up to data cut-off date 09 May 2017 (approximately 15 months)
Population: The analysis population was the FAS.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | ASP8273 | Erlotinib or Gefitinib
Number analyzed (Participants) | 267 | 263
months | 7.43 [5.49 to 9.26] | 10.12 [9.03 to NA] — Data could not be calculated due to low number of events.
Statistical Analysis 1: Comparison: ASP8273 vs Erlotinib or Gefitinib; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.998, Log Rank; Hazard Ratio (HR) = 1.674, 95% CI 2-sided [1.165 to 2.406]

5. Secondary Outcome: Percentage of Participants With Disease Control
Description: Percentage of participants with disease control was defined as the proportion of participants whose best overall response was rated as CR, PR or stable disease (SD) among all analyzed participants based on RECIST V1.1. CR was defined as disappearance of all target and nontarget lesions. Any pathological lymph nodes (whether target or nontarget) must have reduction in short axis to < 10 mm from baseline measurement. PR was defined as at least a 30% decrease in the sum of diameters (longest for nonnodal lesions, short axis for nodal lesions) of target lesions taking as reference to the baseline sum of diameters. SD was defined as neither sufficient decrease to qualify for PR nor sufficient increase to qualify for progressive disease taking as reference the smallest sum of diameters while on study drug.
Time Frame: From date of first dose of study drug up to data cut-off date 09 May 2017 (approximately 15 months)
Population: The analysis population was the FAS.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | ASP8273 | Erlotinib or Gefitinib
Number analyzed (Participants) | 267 | 263
percentage of participants | 62.2 [56.1 to 68.0] | 66.2 [60.1 to 71.9]
Statistical Analysis 1: Comparison: ASP8273 vs Erlotinib or Gefitinib; [analysis description as in outcome 3, analysis 1]; Test type: Superiority; p = 0.839, Cochran-Mantel-Haenszel

6. Secondary Outcome: Duration of Response (DOR)
Description: DOR was defined as the time from the date of the first response CR/PR (whichever was first recorded) as assessed by IRR to the date of radiographical progression or date of censoring. If a participant had not progressed, the participant was censored at the date of last radiological assessment or at the date of first CR/PR if no post-baseline radiological assessment was available. Results are based Kaplan-Meier estimate.
Time Frame: From date of first response up to data cut-off date 09 May 2017 (approximately 15 months)
Population: The analysis population was the FAS. Only participants with best overall response as CR or PR (without confirmation) were included in the analysis.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | ASP8273 | Erlotinib or Gefitinib
Number analyzed (Participants) | 88 | 126
months | 9.17 [5.45 to NA] — Data could not be calculated due to low number of events. | 9.03 [7.39 to NA] — Data could not be calculated due to low number of events.
Statistical Analysis 1: Comparison: ASP8273 vs Erlotinib or Gefitinib; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.780, Log Rank; Hazard Ratio (HR) = 1.298, 95% CI 2-sided [0.661 to 2.548]

7. Secondary Outcome: Number of Participants With Adverse Events (AEs)
Description: Safety was assessed by AEs, which included abnormalities identified during a medical test (e.g. laboratory tests, vital signs, electrocardiogram, etc.) if the abnormality induced clinical signs or symptoms, needed active intervention, interruption or discontinuation of study medication or was clinically significant. A treatment-emergent AE (TEAE) was defined as an AE observed after starting administration of the study drug. AEs were considered serious (SAEs) if the AE resulted in death, was life threatening, resulted in persistent or significant disability/incapacity or substantial disruption of the ability to conduct normal life functions, resulted in congenital anomaly, or birth defect or required inpatient hospitalization or led to prolongation of hospitalization.
Time Frame: From first dose of study drug up to 30 days after last dose of study drug taken up to data cut-off 09 May 2017
Population: The analysis population was SAF.
Measure: Number; unit: participants
Arm/Group | ASP8273 | Erlotinib or Gefitinib
Number analyzed (Participants) | 265 | 262
participants
  TEAE | 251 | 261
  Drug-Related TEAE | 235 | 246
  Serious TEAE | 84 | 67
  Drug-Related Serious TEAE | 46 | 18
  TEAE Leading to Death | 14 | 17
  Drug-Related TEAE Leading to Death | 1 | 1
  TEAE Leading to Treatment Withdrawal | 39 | 28
  Drug-Related TEAE Leading to Treatment Withdrawal | 27 | 17
  TEAE Leading to Dose Reduction | 51 | 51
  Drug-Related TEAE Leading to Dose Reduction | 51 | 50
  TEAE Leading to Dose Interruption | 95 | 74
  Drug-Related TEAE Leading to Dose Interruption | 83 | 55
  Death | 39 | 35

8. Secondary Outcome: Functional Assessment of Cancer Therapy - EGFR Inhibitors Subscale (FACT-EGFRI-18) Questionnaire
Description: ACT-EGFRI-18 is an 18-item Likert-scaled questionnaire, used to assess the effect of EGFR inhibitors on quality of life (QoL). The questionnaire is arranged in three HRQL dimensions: physical (seven items), social/emotional (six items), and functional well-being (five items). The response scores ranged from 0 to 4, and the response categories include "not at all", "a little bit", "somewhat", "quite a bit", and "very much." Negatively worded items (e.g., "My skin bleeds easily "or "My skin condition affects my mood") are reverse-scored, so that participants who experience a higher impact of symptom burden on HRQL receive a lower score (range 0-72).
Time Frame: Day 1 of each cycle up to data cut off 09 May 2017 (approximately 15 months)
Population: The analysis population was the SAF, with available data.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | ASP8273 | Erlotinib or Gefitinib
Number analyzed (Participants) | 248 | 251
units on a scale | 2.79 (4.97) | 9.34 (10.57)

9. Secondary Outcome: European Organisation for Research and Treatment of Cancer Quality of Life Questionnaire - Lung Cancer 13 (EORTC-QLQ-LC13)
Description: The EORTC-QLQ-LC13 is a validated module of the EORTC-QLQ-Core 30, which includes module items that evaluate symptoms such as cough, hemoptysis, shortness of breath, sore mouth or tongue, dysphagia, tingling hands or feet, hair loss and pain. The total score for the questionnaire ranges from 0 to 100. A high score for a functional scale represents a high/healthy level of functioning whereas a high score for a symptom scale or item represents a high level of symptomatology or problems.
Time Frame: Day 1 of each cycle up to data cut off 09 May 2017 (approximately 15 months)
Population: The analysis population was the SAF, with available data.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | ASP8273 | Erlotinib or Gefitinib
Number analyzed (Participants) | 248 | 251
units on a scale | 18.93 (4.42) | 18.78 (4.69)

10. Secondary Outcome: European Organisation for Research and Treatment of Cancer Core Quality of Life Questionnaire (EORTC-QLQ-C30)
Description: EORTC-QLQ-LC30 is a 30-item cancer-specific questionnaire with multitrait scaling was used to create five functional domain scales: Physical, Role, Emotional, Social and Cognitive; two items evaluate global QoL; in addition, three symptom scales assess Fatigue, Pain and Emesis; and six single items assess other symptoms. The total score ranges from 0 to 100, with a high score for a functional scale representing a high/healthy level of functioning and a high score for a symptom scale or item representing a high level of symptomatology or problems.
Time Frame: Day 1 of each cycle up to data cut off 09 May 2017 (approximately 15 months)
Population: The analysis population was the SAF, with available data.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | ASP8273 | Erlotinib or Gefitinib
Number analyzed (Participants) | 248 | 251
units on a scale | 53.77 (11.49) | 52.01 (11.26)

11. Secondary Outcome: EuroQol 5-Dimension 5-Level Questionnaire (EQ-5D-5L)
Description: The EQ-5D is a generic preference-based measure that indirectly measures the utility for health that generates an index-based summary score based upon societal preference weights. The EQ-5D-5L consists of 6 items that cover 5 main domains (mobility, self-care, usual activities, pain/discomfort, and anxiety/depression) and a general visual analog scale (VAS) for health status. Each item has 5 response levels ranging from level 1 (no problem or none) to level 5 (unable to perform activity). The VAS ranges from 0 (worst health status) and 100 (best health status).
Time Frame: Day 1 of each cycle up to data cut off 09 May 2017 (approximately 15 months)
Population: The analysis population was the SAF, with available data.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | ASP8273 | Erlotinib or Gefitinib
Number analyzed (Participants) | 248 | 251
Units on a scale
  Mobility | 1.78 (0.96) | 1.48 (0.85)
  Self-care | 1.28 (0.68) | 1.19 (0.60)
  Usual Activities | 1.71 (0.94) | 1.54 (0.83)
  Pain/Discomfort | 1.79 (0.86) | 1.71 (0.83)
  Anxiety/Depression | 1.61 (0.77) | 1.54 (0.76)
  VAS | 69.44 (19.17) | 72.36 (17.19)

ADVERSE EVENTS:
Time Frame: From first dose of study drug up to 30 days after last dose of study drug taken up to data cut-off 21 Dec 2017 (approximately 22 months)
Arm/Group | ASP8273 | Erlotinib or Gefitinib
All-Cause Mortality (participants affected / at risk) | 39/265 | 35/262
Serious Adverse Events (participants affected / at risk) | 84/265 | 67/262
Other Adverse Events (participants affected / at risk) | 240/265 | 253/262
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ASP8273 (N=265) | Erlotinib or Gefitinib (N=262)
Anaemia (Blood and lymphatic system disorders) | 2 (2) | 0 (0)
Acute myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0)
Angina pectoris (Cardiac disorders) | 1 (1) | 0 (0)
Atrial thrombosis (Cardiac disorders) | 0 (0) | 1 (1)
Pericardial effusion (Cardiac disorders) | 0 (0) | 2 (3)
Deafness unilateral (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Retinal artery occlusion (Eye disorders) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 2 (2) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1) | 0 (0)
Colitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 7 (7) | 2 (2)
Enterocolitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastritis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 (1) | 0 (0)
Intussusception (Gastrointestinal disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 2 (2) | 0 (0)
Oesophagitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Pancreatitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Umbilical hernia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 2 (2) | 0 (0)
Vomiting (Gastrointestinal disorders) | 3 (3) | 0 (0)
Asthenia (General disorders) | 2 (2) | 1 (1)
Chest pain (General disorders) | 1 (1) | 0 (0)
Death (General disorders) | 1 (1) | 0 (0)
Fatigue (General disorders) | 2 (2) | 0 (0)
Gait disturbance (General disorders) | 1 (1) | 0 (0)
Non-cardiac chest pain (General disorders) | 1 (2) | 0 (0)
Pyrexia (General disorders) | 3 (3) | 1 (1)
Biliary colic (Hepatobiliary disorders) | 0 (0) | 1 (1)
Drug-induced liver injury (Hepatobiliary disorders) | 1 (2) | 0 (0)
Hepatic failure (Hepatobiliary disorders) | 1 (1) | 0 (0)
Hepatic function abnormal (Hepatobiliary disorders) | 0 (0) | 1 (1)
Bacteraemia (Infections and infestations) | 0 (0) | 1 (1)
Bronchitis (Infections and infestations) | 1 (1) | 0 (0)
Bronchopneumonia (Infections and infestations) | 0 (0) | 1 (1)
Cellulitis (Infections and infestations) | 0 (0) | 3 (5)
Dengue fever (Infections and infestations) | 1 (1) | 0 (0)
Diarrhoea infectious (Infections and infestations) | 0 (0) | 1 (1)
Escherichia urinary tract infection (Infections and infestations) | 2 (2) | 0 (0)
Influenza (Infections and infestations) | 1 (1) | 0 (0)
Lung infection (Infections and infestations) | 2 (3) | 1 (1)
Pneumonia (Infections and infestations) | 11 (15) | 5 (5)
Pulmonary tuberculosis (Infections and infestations) | 0 (0) | 1 (1)
Sepsis (Infections and infestations) | 3 (3) | 1 (1)
Septic shock (Infections and infestations) | 2 (3) | 1 (1)
Soft tissue infection (Infections and infestations) | 0 (0) | 1 (1)
Staphylococcal bacteraemia (Infections and infestations) | 0 (0) | 1 (1)
Superinfection fungal (Infections and infestations) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (2) | 1 (1)
Urinary tract infection bacterial (Infections and infestations) | 1 (1) | 0 (0)
Urinary tract infection enterococcal (Infections and infestations) | 0 (0) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Femoral neck fracture (Injury, poisoning and procedural complications) | 2 (3) | 0 (0)
Femur fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Procedural nausea (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Procedural pain (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Radius fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Alanine aminotransferase increased (Investigations) | 1 (1) | 3 (9)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 2 (6)
Blood alkaline phosphatase increased (Investigations) | 0 (0) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 3 (3) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Diabetes mellitus (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypoglycaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 2 (2) | 1 (1)
Hyponatraemia (Metabolism and nutrition disorders) | 14 (17) | 1 (1)
Arthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 3 (3)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Acute myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (3)
Bowen's disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (2)
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 6 (7) | 8 (9)
Malignant pleural effusion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0)
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 2 (2)
Metastases to eye (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Metastases to meninges (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (3) | 1 (1)
Neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (2) | 0 (0)
Neoplasm skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (2)
Tumour haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0)
Altered state of consciousness (Nervous system disorders) | 1 (1) | 0 (0)
Aphasia (Nervous system disorders) | 1 (1) | 0 (0)
Brain oedema (Nervous system disorders) | 1 (2) | 0 (0)
Depressed level of consciousness (Nervous system disorders) | 1 (1) | 0 (0)
Dysarthria (Nervous system disorders) | 1 (1) | 0 (0)
Embolic stroke (Nervous system disorders) | 1 (1) | 0 (0)
Encephalopathy (Nervous system disorders) | 1 (2) | 0 (0)
Epilepsy (Nervous system disorders) | 0 (0) | 1 (1)
Haemorrhage intracranial (Nervous system disorders) | 1 (2) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 1 (1)
Paraesthesia (Nervous system disorders) | 1 (1) | 0 (0)
Partial seizures (Nervous system disorders) | 0 (0) | 1 (1)
Peripheral sensory neuropathy (Nervous system disorders) | 1 (1) | 0 (0)
Seizure (Nervous system disorders) | 2 (2) | 0 (0)
Spinal cord compression (Nervous system disorders) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 1 (1) | 0 (0)
Agitation (Psychiatric disorders) | 1 (1) | 0 (0)
Confusional state (Psychiatric disorders) | 1 (1) | 0 (0)
Delirium (Psychiatric disorders) | 1 (1) | 0 (0)
Depression (Psychiatric disorders) | 1 (1) | 0 (0)
Mental status changes (Psychiatric disorders) | 1 (2) | 1 (1)
Psychotic disorder (Psychiatric disorders) | 1 (1) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 5 (5) | 2 (3)
Chronic kidney disease (Renal and urinary disorders) | 1 (1) | 0 (0)
Haematuria (Renal and urinary disorders) | 1 (1) | 0 (0)
Renal impairment (Renal and urinary disorders) | 0 (0) | 1 (1)
Urinary retention (Renal and urinary disorders) | 1 (1) | 0 (0)
Prostatitis (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (3)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 5 (6) | 3 (4)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 3 (5)
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 4 (7)
Pharyngeal inflammation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (2)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 1 (1)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (6)
Drug eruption (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2)
Hypertension (Vascular disorders) | 1 (1) | 0 (0)
Hypertensive crisis (Vascular disorders) | 0 (0) | 1 (1)
Hypotension (Vascular disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ASP8273 (N=265) | Erlotinib or Gefitinib (N=262)
Anaemia (Blood and lymphatic system disorders) | 21 (27) | 17 (30)
Dry eye (Eye disorders) | 7 (8) | 17 (21)
Constipation (Gastrointestinal disorders) | 54 (68) | 24 (24)
Diarrhoea (Gastrointestinal disorders) | 161 (255) | 135 (224)
Dry mouth (Gastrointestinal disorders) | 30 (31) | 1 (1)
Nausea (Gastrointestinal disorders) | 66 (85) | 33 (41)
Stomatitis (Gastrointestinal disorders) | 18 (21) | 55 (70)
Vomiting (Gastrointestinal disorders) | 51 (60) | 26 (31)
Asthenia (General disorders) | 31 (39) | 19 (28)
Fatigue (General disorders) | 50 (73) | 30 (47)
Pyrexia (General disorders) | 18 (22) | 17 (20)
Paronychia (Infections and infestations) | 5 (6) | 67 (106)
Upper respiratory tract infection (Infections and infestations) | 10 (11) | 18 (24)
Alanine aminotransferase increased (Investigations) | 53 (125) | 51 (107)
Aspartate aminotransferase increased (Investigations) | 36 (67) | 43 (88)
Blood bilirubin increased (Investigations) | 4 (4) | 15 (28)
Platelet count decreased (Investigations) | 18 (25) | 3 (5)
Weight decreased (Investigations) | 17 (17) | 21 (27)
Decreased appetite (Metabolism and nutrition disorders) | 56 (73) | 48 (64)
Hyponatraemia (Metabolism and nutrition disorders) | 64 (134) | 7 (13)
Arthralgia (Musculoskeletal and connective tissue disorders) | 14 (16) | 7 (7)
Back pain (Musculoskeletal and connective tissue disorders) | 14 (16) | 18 (22)
Dizziness (Nervous system disorders) | 29 (29) | 11 (11)
Dysgeusia (Nervous system disorders) | 30 (35) | 10 (10)
Headache (Nervous system disorders) | 21 (25) | 23 (25)
Paraesthesia (Nervous system disorders) | 19 (22) | 7 (7)
Peripheral sensory neuropathy (Nervous system disorders) | 57 (76) | 2 (2)
Insomnia (Psychiatric disorders) | 22 (24) | 17 (17)
Cough (Respiratory, thoracic and mediastinal disorders) | 25 (28) | 30 (41)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 20 (25) | 16 (16)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 6 (6) | 15 (15)
Alopecia (Skin and subcutaneous tissue disorders) | 8 (8) | 37 (42)
Drug eruption (Skin and subcutaneous tissue disorders) | 32 (34) | 186 (377)
Dry skin (Skin and subcutaneous tissue disorders) | 32 (33) | 66 (83)
Pruritus (Skin and subcutaneous tissue disorders) | 12 (13) | 35 (44)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Institute and/or Principal Investigator may publish trial data generated at their specific study site after Sponsor publication of the muli-center data. Sponsor must receive a site's manuscript prior to publication for review and comment as specified in the Investigator Agreement.

DOCUMENTS (2):
  • Study Protocol (2016-02-19): https://cdn.clinicaltrials.gov/large-docs/61/NCT02588261/Prot_000.pdf
  • Statistical Analysis Plan (2016-08-11): https://cdn.clinicaltrials.gov/large-docs/61/NCT02588261/SAP_001.pdf